CLINICAL TRIAL: NCT06623539
Title: Pemafibrate for Treating NAFLD Complicated by Hypertriglyceridemia: A Multi-center, Open Study, Randomized Controlled Trial (PRESENT Study)
Brief Title: Efficacy and Safety of Pemafibrate for Nonalcoholic Fatty Liver Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yokohama City University (Other)
Responsible Party: Principal Investigator, Hidenori Ohkubo, Michihiro Iwaki, Yokohama City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jRCTs031200280
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Pemafibrate; Fenofibrate
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid; Fenofibrate

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, three-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pemafibrate high dose group (Experimental)
  Interventions: Drug: Pemafibrate high dose
- Pemafibrate low dose group (Experimental)
  Interventions: Drug: Pemafibrate low dose
- Fenofibrate group (Experimental)
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Pemafibrate high dose — Pemafibrate 0.1 mg tablets shall be administered orally twice daily, two tablets per dose, after the morning and evening meals. If unavoidable, pemafibrate extended-release 0.2 mg for 2 tablets 1 or 0.4 mg for 1 tablet 1 can be substituted.
  Arms: Pemafibrate high dose group
Drug: Pemafibrate low dose — Pemafibrate 0.1 mg tablets shall be administered orally twice daily, one tablet per dose, after the morning and evening meals. If unavoidable, pemafibrate extended-release 0.2 mg for 1 tablets 1 can be substituted.
  Arms: Pemafibrate low dose group
Drug: Fenofibrate — Fenofibrate 53.3 mg tablets shall be administered orally once daily, one tablet per dose, after breakfast. Thereafter, the dose may be carefully increased to two tablets per dose at the physician's discretion.
  Arms: Fenofibrate group

SUMMARY:
This is a study to evaluate the effect of pemafibrate on fatty liver in patients with hypertgemia combined with NAFLD, using fenofibrate as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 20 years old and under 80 years old at the time of obtaining consent.
2. Patients with fatty liver diagnosed histologically within 1 year prior to obtaining consent or imaging examination within 6 months prior to obtaining consent and who have failed exercise and diet therapy for at least 3 months.
3. Patients with hypertriglyceridemia (150-500 mg/dl) within 91 days prior to obtaining consent.
4. Patients with elevated ALT (43-100 IU/L for men, 24-100 IU/L for women) within 91 days prior to obtaining consent.
5. Patients whose daily alcohol consumption (ethanol equivalent) is less than 30 grams per day for men and less than 20 grams per day for women at the time of obtaining consent.
6. Patients with hepatitis C, hepatitis B (excluding inactive carriers), autoimmune hepatitis, primary biliary cholangitis, or other hepatic complications that have been ruled out at the time of obtaining consent.
7. Patients whose written consent to participate in this study has been obtained. [Basis for settings]

1） The age range was set to 20 years or older because the safety of the study drug has not been established in children. In addition, the age of patients was set to be less than 80 years considering safety and the susceptible age of NAFLD/NASH onset.

2） This is because the 2014 NAFLD/NASH guideline states that "fatty liver is present on histology or imaging" regarding NAFLD definition.

3） Within dyslipidemia patients, those with hypertriglyceridemia and indicated for fibrates will be used as controls.

Since TG>500 poses a risk of developing acute pancreatitis, the selection criteria were TG levels between 150 and 500 mg/dl.

4） Since the primary endpoint in this study was the amount of change in ALT, elevated ALT was used as the selection criterion in the JCCLS shared reference value range so that changes could be better understood. ALT was specifically set as the upper limit of normal to 100 IU/L in the selection criteria based on the package insert of fenofibrate.

5） NAFLD diagnostic criteria from the 2014 NAFLD/NASH guidelines were cited. 6） NAFLD diagnostic criteria from the 2014 NAFLD/NASH guidelines were cited. 7） This was set to ensure the free and voluntary participation of the study participants.

Exclusion Criteria:

1. Patients taking contraindications (see "6.5.2.2 Contraindicated treatments").

   Cyclosporine, rifampicin, steroids (excluding topical and inhaled drugs), amiodarone, breast cancer drugs (tamoxifen, toremifene, raloxifene).
2. Patients with BMI <18.5 kg/m2 at the time of obtaining consent.
3. Patients who have been diagnosed with liver cirrhosis at the time of obtaining consent.
4. Patients with findings of portal hypertension (varicose veins, ascites, encephalopathy, splenomegaly) at the time of obtaining consent.
5. Patients with T-Bil > 2× the upper limit of normal within 91 days prior to obtaining consent, excluding Girbert syndrome.
6. Platelet count <80,000/μL within 91 days prior to obtaining consent.
7. Serum Cr level of 1.5 mg/dL or higher within 91 days prior to obtaining consent.
8. Patients with gallstones or biliary obstruction at the time of obtaining consent.
9. Patients with severe infection, pre- or post-operative, or severe trauma at the time of obtaining consent.
10. Patients who have used fibrates within 91 days prior to obtaining consent
11. Patients with 10% weight change in 91 days prior to obtaining consent
12. Patients who have undergone bariatric surgery or are scheduled for surgery during the study period
13. Patients with a history of type I diabetes mellitus
14. Patients with HbA1c >9.5% within 91 days prior to obtaining consent (If HbA1c >9.5%, re-entry will be possible after improvement by treatment.)
15. Patients with psychosis, alcoholism, drug addiction, or narcotic addiction that would affect compliance with the research protocol
16. Patients who participated in other clinical trials in 100 days prior to obtaining consent
17. Pregnant women or patients who may be pregnant
18. Patients with complications of malignant tumors However, patients who have undergone radical surgery or completed anticancer drug administration may enroll. Patients under observation and evaluation for malignant tumors are excluded.
19. Other patients who are judged by the investigator to be inappropriate as participants of this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in ALT level | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yokohama city university, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No